CLINICAL TRIAL: NCT07057713
Title: A Prospective, Randomized, Double-Blind Controlled Trial Comparing Total Arterial Grafting Versus Conventional Mixed Grafting in the Left Coronary Artery System During Coronary Artery Bypass Grafting (CABG)
Brief Title: Total Arterial vs. Mixed Grafting in Left Coronary CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kexiang Liu, MD, Principal Investigator, Second Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDEYXWK208
Record Dates: First submitted 2025-06-29; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting; Arterial Graft; Graft Patency; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients undergoing elective CABG will be randomized 1:1 to receive either total arterial grafting or conventional mixed grafting in the left coronary system.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blinded to the grafting strategy. The surgical team will not be blinded due to the nature of the intervention, but outcome evaluation will be conducted by independent, blinded assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Arterial Grafting Group (Experimental): Patients in this group will undergo coronary artery bypass grafting (CABG) with total arterial grafts to the left coronary artery system. The left internal thoracic artery (LITA) will be grafted to the left anterior descending artery (LAD), and the radial artery will be anastomosed to the obtuse marginal or diagonal branches of the circumflex artery. The right coronary artery, if revascularized, will receive a conventional vein graft.
  Interventions: Procedure: Total Arterial Grafting
- Conventional Mixed Grafting Group (Active Comparator): Patients in this group will receive conventional mixed grafting during CABG. The left internal thoracic artery (LITA) will be used for the LAD, while the great saphenous vein will be grafted to other branches of the left coronary artery system, such as the obtuse marginal or diagonal branches. The right coronary artery, if revascularized, will also be grafted using a vein.
  Interventions: Procedure: Conventional Mixed Grafting

INTERVENTIONS:
Procedure: Total Arterial Grafting — Coronary artery bypass grafting using only arterial conduits in the left coronary artery system. The left internal thoracic artery (LITA) is grafted to the LAD, and the radial artery is anastomosed to the obtuse marginal or diagonal branches. This approach avoids the use of saphenous vein grafts for the left coronary system.
  Other Names: LITA + Radial Artery Grafting
  Arms: Total Arterial Grafting Group
Procedure: Conventional Mixed Grafting — A standard coronary artery bypass grafting (CABG) procedure where the left internal thoracic artery (LITA) is grafted to the LAD, and saphenous vein grafts are used for the obtuse marginal or diagonal branches of the left coronary system. This approach represents the conventional mixed arterial-venous strategy.
  Other Names: Mixed Arterial-Venous Grafting
  Arms: Conventional Mixed Grafting Group

SUMMARY:
This is a prospective, randomized, double-blind controlled trial comparing the clinical efficacy of total arterial grafting (internal thoracic artery and radial artery) versus conventional mixed grafting (internal thoracic artery and great saphenous vein) in the left coronary artery system during coronary artery bypass grafting (CABG). A total of 400 patients undergoing elective CABG at the Second Hospital of Jilin University will be enrolled and randomized into two groups. The primary endpoint is graft patency at 12 months postoperatively, evaluated by coronary angiography or CT angiography. Secondary outcomes include perioperative complications, major adverse cardiovascular events (MACE), and long-term clinical prognosis. The study aims to provide evidence-based guidance on optimal graft selection in CABG.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) remains a cornerstone treatment for multivessel coronary artery disease. The choice of conduit significantly affects long-term graft patency and patient outcomes. While the left internal thoracic artery (LITA) to the left anterior descending artery (LAD) is standard, the optimal strategy for other coronary territories-such as the circumflex and right coronary arteries-remains debated.

This prospective, randomized, double-blind controlled trial aims to evaluate the long-term clinical efficacy of total arterial grafting (LITA + radial artery) versus conventional mixed grafting (LITA + great saphenous vein) in the left coronary artery system. A total of 400 patients scheduled for elective CABG at the Second Hospital of Jilin University will be enrolled and randomly assigned to one of the two surgical strategies. The experimental group will receive total arterial grafts to the LAD and circumflex branches, while the control group will receive arterial graft to LAD and vein grafts to the circumflex.

The primary endpoint is graft patency at 12 months post-surgery, assessed via coronary angiography or CT angiography. Secondary outcomes include major adverse cardiovascular events (MACE), perioperative complications (e.g., myocardial infarction, atrial fibrillation, infection), and long-term changes in cardiac function (e.g., LVEF, NYHA class). All surgeries will be performed by the same experienced surgical team following standardized procedures.

Patients will be followed at 1, 6, and 12 months postoperatively. Data will be collected through the hospital electronic medical record system and analyzed with appropriate statistical methods, including Cox proportional hazards modeling and Kaplan-Meier survival curves. Ethical approval has been obtained, and informed consent will be required from all participants. This study is designed to provide high-level evidence to optimize graft selection strategies in CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosed with multivessel coronary artery disease
3. Indicated for elective coronary artery bypass grafting (CABG) involving ≥3 coronary vessels
4. Right coronary artery stenosis >75%
5. Able and willing to provide written informed consent

Exclusion Criteria:

1. Scheduled for concurrent cardiac procedures (e.g., valve surgery, congenital heart disease repair, aortic dissection surgery, atrial fibrillation ablation)
2. Severe stenosis of left or right subclavian artery
3. Unsuitable saphenous veins (e.g., bilateral varicosities)
4. Unsuitable radial artery as assessed preoperatively
5. History of intracranial hemorrhage or ischemic stroke within the past 14 days
6. Severe hepatic or renal insufficiency
7. Acute myocardial infarction within 72 hours prior to surgery
8. History of prior CABG or other cardiac surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Graft Patency Rate | 12 months after surgery
  Graft patency will be assessed at 12 months after surgery by coronary angiography or coronary CT angiography. A patent graft is defined as one with <50% stenosis and continuous flow. The proportion of patients with all coronary artery grafts remaining patent will be calculated and compared between groups.

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events | Within 12 months after surgery
  MACE includes cardiac death, nonfatal myocardial infarction, and the need for repeat revascularization. Events will be recorded during hospitalization and follow-up visits up to 12 months after surgery.
Incidence of Perioperative Complications | Within 30 days after surgery
  Includes postoperative atrial fibrillation, stroke, wound infection, renal insufficiency, and reoperation for bleeding. Data will be collected during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Kexiang Liu, Principal Investigator — Department of Cardiovascular Surgery, The Second Hospital of Jilin University
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No